CLINICAL TRIAL: NCT06223854
Title: Evaluation of the Acceptability and Nutritional Effects of Double-fortified Salt Containing Folic Acid and Iodine Among Ethiopian Women of Reproductive Age - a Household-randomized, Controlled, Community-based Trial
Brief Title: Acceptability and Nutritional Impact of Double-fortified Salt Containing Iodine and Folic Acid
Acronym: DFS-IoFA-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Ethiopian Public Health Institute (Other Government); University of California, San Francisco (Other); University of Rhode Island (Other); Nutrition International (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2078626
Record Dates: First submitted 2024-01-03; First posted 2024-01-25 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-01

CONDITIONS: Folate Deficiency; Iodine Deficiency; Anemia Macrocytic; Anemia Deficiency; Salt Intake; Vitamin B 12 Deficiency
Keywords: Salt fortification; Ethiopia
MeSH Terms: conditions — Folic Acid Deficiency; Anemia, Macrocytic; Vitamin B 12 Deficiency | interventions — iodized salt

STUDY DESIGN:
Intervention Model Description: This study is a community-based, three-arm, randomized, dose-response intervention trial with randomization at the level of the household of non-pregnant women of reproductive age.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The salts will be packaged in 500-gram plastic containers (canisters) labeled with the participants' study identification number. Two containers of salt will be delivered to the participants' homes every two weeks, at which time the previously delivered canisters will be collected..
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Iodized salt (Active Comparator): Refined iodized salt containing 35 ppm iodine as potassium iodate
  Interventions: Dietary Supplement: Iodized salt
- Iodized salt with lower-dose folic acid fortification (Experimental): Refined iodized salt containing 35 ppm iodine as potassium iodate and 33 ppm folic acid (to provide an estimated 200 microgram folic acid per day to women consuming the previously determined average amount of discretionary salt in the study communities)
  Interventions: Dietary Supplement: Experimental: Iodized salt with lower-dose folic acid fortification
- Iodized salt with higher-dose folic acid fortification (Experimental): Refined iodized salt containing 35 ppm iodine as potassium iodate and 99 ppm folic acid (to provide an estimated 600 microgram folic acid per day to women consuming the previously average amount of discretionary salt in the study communities)
  Interventions: Dietary Supplement: Experimental: Iodized salt with higher-dose folic acid fortification

INTERVENTIONS:
Dietary Supplement: Iodized salt — Masked, individually labeled 500-g containers of the study salts will be delivered to the participants' homes bi-weekly by field workers who will collect previously delivered salt containers during the same visit. Participants will be counseled to use the study salt for all food preparation and meal-time seasoning for all members of the household and not to share the salt with others or use it for non-food consumption purposes.
  Arms: Iodized salt
Dietary Supplement: Experimental: Iodized salt with lower-dose folic acid fortification — Masked, individually labeled 500-g containers of the study salts will be delivered to the participants' homes bi-weekly by field workers who will collect previously delivered salt containers during the same visit. Participants will be counseled to use the study salt for all food preparation and meal-time seasoning for all members of the household and not to share the salt with others or use it for non-food consumption purposes.
  Arms: Iodized salt with lower-dose folic acid fortification
Dietary Supplement: Experimental: Iodized salt with higher-dose folic acid fortification — Masked, individually labeled 500-g containers of the study salts will be delivered to the participants' homes bi-weekly by field workers who will collect previously delivered salt containers during the same visit. Participants will be counseled to use the study salt for all food preparation and meal-time seasoning for all members of the household and not to share the salt with others or use it for non-food consumption purposes.
  Arms: Iodized salt with higher-dose folic acid fortification

SUMMARY:
The overarching objective of this two-phase project is to assess the effects of fortifying iodized salt with folic acid on improving women's folate status. Folate insufficiency is the primary risk factor for neural tube defects (NTDs), which are highly prevalent in Ethiopia. The purposes of Phase 2 of the project, described herein, are to complete a community-based, randomized, dose-response intervention trial of edible salt fortified with just iodine or iodine and one of two levels of folic acid among non-pregnant women of reproductive age (WRA), We will assess the effects of the intervention on women's discretionary salt intakes, markers of folate and iodine status, and incidence of any adverse events.

DETAILED DESCRIPTION:
Potentially eligible women of reproductive age (WRA) in two rural and two semi-urban communities (kebeles) in the Oromia Region of Ethiopia will be identified from existing census records. A convenience sample of 360 eligible, consenting women will be recruited following an initial screening interview at the women's homes. Before the screening interview, the data collector will read a disclosure statement concerning the purpose and the contents of the interview, and the data collector will then request verbal consent to obtain descriptive information on the women's age, general health status, pregnancy status, use of contraceptives, address, cell phone number (if available), and potential willingness to participate in the subsequent intervention trial.

After reviewing the women's health history and pregnancy status, measured blood pressure, and current use of contraceptives, the data collector will determine the women's potential eligibility for the trial. The data collector will describe the purposes of the trial, the study procedures and related risks and benefits, the confidentiality of results, and the fact that participation is voluntary. Women who are interested in participating in the study will be encouraged to ask any questions to the research team and consult with family members before providing their signed consent (in the presence of a neutral witness) to participate in the trial. Additional questions then will be asked of consenting women regarding their marital status, ethnicity, religion, educational level, and employment; and their housing characteristics (housing construction, water source, sanitary facilities, access to electricity and cell phone service), and selected household (HH) assets; and the women will be invited to attend the local health facility to complete additional interviews to assess their birth history, household food insecurity, and additional eligibility criteria, including anthropometrics, a pregnancy test, and fasting blood collection for anemia screening and other baseline measurements. Eligible, consenting women then will be randomly assigned to one of three study arms using a block randomization procedure with block size of six. The fasting blood samples obtained for anemia screening will also be used for measurement of red blood cell and serum folate, unmetabolized folic acid, homocysteine, vitamin B12, holo-transcobalamin, methyl malonic acid, other B vitamins, genetic polymorphisms that affect folate metabolism, thyroglobulin, glucose, insulin, retinol binding protein (RBP), ferritin, soluble transferrin receptor, C-reactive protein, and alpha-1 acid glycoprotein, and a malaria rapid diagnostic test (RDT).

Following enrollment, the study participants will be scheduled for a 24-hour urine collection to measure baseline sodium and iodine excretion, after which they will begin receiving the assigned study salt every two weeks. The women will be counseled to use the study salt for all food preparation and seasoning for a total of 26 weeks. Additional data collection during the course of the intervention will include: one or two full-day observed food records to measure discretionary salt intake and folate intake; one or two repeat 24-hour urine collections to measure sodium and iodine excretion; and bi-weekly home assessments of salt acceptability, continued contraceptive use, and any adverse events. At the time of these bi-weekly home visits, unused salt will be collected and a new allotment of salt will be delivered. Fasting blood samples will be collected again at a randomly assigned intermediate time point and at end line.

- Page 2 of 5 -

ELIGIBILITY:
Inclusion Criteria:

* Non-pregnant
* Using long-acting contraceptive
* Intending to remain in study community for at least six months
* Willing to use study salt for all household food preparation and seasoning
* Signed, informed consent

Exclusion Criteria:

* Pregnant
* Not using long-acting contraceptive
* Acute or chronic disease that affects dietary intake or folate metabolism
* Hypertension
* Medications that potentially interfere with folate metabolism
* Folic acid-containing vitamin supplements
* Macrocytic anemia or moderate/severe non-macrocytic anemia.
* Mid-upper arm circumference <23 cm and breast feeding an infant <6 months of age

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 360 (Actual)
Dates: Start 2024-04-25 (Actual); Primary Completion 2024-12-16 (Actual); Study Completion 2024-12-16 (Actual)

PRIMARY OUTCOMES:
Red blood cell folate | Baseline (pre-intervention), intermediate time point (between 4-20 weeks), and end line (24-26 weeks)
  Red blood cell (RBC) folate concentration will be measured on three occasions in each participant: 1) before the start of the intervention, 2) at a randomly assigned mid-point between 4 and 20 weeks after the start of the intervention, and 3) between 24-26 weeks after the start of the intervention. RBC folate concentration will be will be determined by using a microbiological assay.
Serum folate | Baseline (pre-intervention), intermediate time point (between 4-20 weeks), and end line (24-26 weeks)
  Serum folate concentration will be measured on three occasions in each participant: 1) before the start of the intervention, 2) at a randomly assigned mid-point between 4 and 20 weeks after the start of the intervention, and 3) between 24-26 weeks after the start of the intervention, by using a microbiological assay.
Serum homocysteine | Baseline (pre-intervention), intermediate time point (between 4-20 weeks), and end line (24-26 weeks)
  Serum homocysteine concentration will be measured on three occasions in each participant: 1) before the start of the intervention, 2) at a randomly assigned mid-point between 4 and 20 weeks after the start of the intervention, and 3) between 24-26 weeks after the start of the intervention.
Serum thyroglobulin | Baseline (pre-intervention), intermediate time point (between 4-20 weeks), and end line (24-26 weeks)
  Serum thyroglobulin concentration will be measured on three occasions in each participant: 1) before the start of the intervention, 2) at a randomly assigned mid-point between 4 and 20 weeks after the start of the intervention, and 3) between 24-26 weeks after the start of the intervention.
24-hour urinary iodine excretion | Before and during the intervention
  24-hour urinary iodine excretion will be measured prior to the start of the intervention and at a second time time at least 4 weeks after the start of the intervention.
Serious adverse events | Throughout the course of the intervention, total of 26 weeks
  Serious adverse events requiring an overnight stay in a clinical facility or resulting in disability, or death will be recorded during each bi-weekly home visit.

SECONDARY OUTCOMES:
Hemoglobin concentration | Baseline (pre-intervention), intermediate time point (between 4-20 weeks), and end line (24-26 weeks)
  Hemoglobin concentration in venous blood will be measured at three time points, using an automated hematology analyzer.
Serum B12 | Baseline (pre-intervention), intermediate time point (between 4-20 weeks), and end line (24-26 weeks)
  Serum concentration of cyanocobalamin will be measured at three time points.
Serum transcobalamin | Baseline (pre-intervention), intermediate time point (between 4-20 weeks), and end line (24-26 weeks)
  Serum concentration of transcobalamin will be measured at three time points.
Serum methyl malonic acid | Baseline (pre-intervention), intermediate time point (between 4-20 weeks), and end line (24-26 weeks)
  Serum concentration of methyl malonic acid will be measured at three time points.
Serum unmetabolized folic acid | Baseline (pre-intervention), intermediate time point (between 4-20 weeks), and end line (24-26 weeks)
  Unmetabolized folic acid will be measured in serum at three time points.
Serum glucose | Baseline (pre-intervention), intermediate time point (between 4-20 weeks), and end line (24-26 weeks)
  Fasting serum glucose concentration will be measured at three time points.
Serum insulin | Baseline (pre-intervention), intermediate time point (between 4-20 weeks), and end line (24-26 weeks)
  Fasting serum insulin concentration will be measured at three time points.
Discretionary salt intake | After the start of the intervention, between 4-20 weeks
  Discretionary salt intake will be measured by full-day, in-home weighed dietary records at one or two time points after the start of the intervention
Urinary sodium excretion | Before and between 4-20 weeks after the start of the intervention
  24-hour urinary sodium excretion will be measured prior to the start of the intervention and at a second time time at least 4 weeks after the start of the intervention.

OTHER OUTCOMES:
Blood pressure | Baseline (pre-intervention), intermediate time point (between 4-20 weeks), and end line (24-26 weeks)
  Resting systolic and diastolic blood pressure will be measured at baseline and at the time of subsequent blood drawings.

CONTACTS AND LOCATIONS:
Overall Officials: KENNETH H BROWN, MD, Principal Investigator — UC Davis; Masresha Tessema, PhD, Principal Investigator — Ethiopian Public Health Institute
Locations (1):
- Ethiopian Public Health Institute, Addis Ababa, Ethiopia

IPD SHARING:
Plan to Share IPD: Yes
Two years after completion of the data collection, the individual participant data (IPD) data sets will become publicly available to other investigators who have specific research questions that can be addressed by the data and that are not already under analysis by the core research team. Researchers who desire to have access to the clinical specimens will be requested to apply for the specimens and to describe the research question(s) they plan to address.
Supporting Information: Study Protocol, ICF
Time Frame: The study protocol will be submitted for publication prior to initiation of Phase 2. The statistical analysis plan will be publicly available prior to the start of the respective analyses. The informed consent documents will be available (in English and Afaan Oromo) .
Access Criteria: As indicated above.

REFERENCES:
- [Background] Brown KH, Tessema M, McDonald CM, Agbemafle I, Woldeyohannes M, Fereja M, Nane D, Arnold CD, Waka FC, Tesfaye B, Arabi M, Martinez H. Protocol for a community-based, household-randomised, dose-response trial to assess the acceptability, nutritional effects and safety of double-fortified salt containing iodine and folic acid compared with iodised salt among non-pregnant Ethiopian women of reproductive age (DFS-IoFA). BMJ Open. 2024 Oct 29;14(10):e084494. doi: 10.1136/bmjopen-2024-084494. PMID 39477275
- [Derived] Tessema M, Nane D, Woldeyohannes M, Agbemafle I, McDonald CM, Arnold CD, Fereja M, Challa F, Martinez H, Tesfaye B, Tollera G, Arabi M, Brown KH; Collaborating Laboratories. Folic acid fortification of iodized salt improves the folate status of non-pregnant adult Ethiopian females and does not impair their iodine status: a community-based, household-randomized, dose-response trial. Am J Clin Nutr. 2026 Jan 27:101204. doi: 10.1016/j.ajcnut.2026.101204. Online ahead of print. PMID 41611087